CLINICAL TRIAL: NCT04117776
Title: Skin Decolonization of Children Hospitalized in Intensive Care Unit by Daily Toilet : Mild Soap Versus Chlorhexidine Gluconate 2% Pad
Brief Title: Skin Decolonization of Children Hospitalized in Intensive Care Unit
Acronym: DCpedrea
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190298; 2019-A00844-53 (Other: IDRCB number)
Record Dates: First submitted 2019-07-01; First posted 2019-10-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Central Venous Catheter
Keywords: Central venous catheter-related bacteremias; Skin decolonization; Intensive care unit hospitalization
MeSH Terms: interventions — Therapeutic Irrigation; chlorhexidine gluconate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patient benefiting during the same hospitalization of the loss or the gain of a central venous catheter.
  Interventions: Other: Skin microbiological sampling (wash with 2% Chlorhexidine Gluconate); Other: Skin microbiological sampling (wash with mild soap)

INTERVENTIONS:
Other: Skin microbiological sampling (wash with 2% Chlorhexidine Gluconate) — 3 microbiological samples, per application of agar on skin, after 24h of a first wash with 2% Chlorhexidine Gluconate : 1h before the second wash with the same washing product and then 1 to 2 h after, and 20 to 23h after this second wash.
  Other Names: Skin microbiological sampling
Other: Skin microbiological sampling (wash with mild soap) — 3 microbiological samples, per application of agar on skin, after 24h of a first wash with mild soap : 1h before the second wash with the same washing product and then 1 to 2 h after, and 20 to 23h after this second wash.
  Other Names: Skin microbiological sampling

SUMMARY:
The purpose of this study is to evaluate the efficacy and duration of the skin decolonization brought by a daily wash using Chlorhexidine Gluconate 2% pad compared to a standard wash with mild soap in children hospitalized in intensive care unit.

DETAILED DESCRIPTION:
Skin is a major reservoir of pathogenic bacteria and intensive care unit patients are particularly vulnerable to variations in skin colonization and so to infections. These bacterial skin colonizations can contaminate other patients, nursing staff or even samples, but above all they are an endogenous source of infection of material. These bacterial skin colonizations hold therefore a major place in the responsibility of infections associated with care and can potentially affect the length of patient hospitalization. 2% Chlorhexidine Gluconate pads have already demonstrated a real efficacy in the sustainable reduction of central venous catheter-related bacteremias in adults and in children, probably through a reduction of cutaneous microbial colonization. However, this hypothesis remains to be confirmed.

Patients in the pediatric surgical intensive care unit of Necker-Enfants Malades hospital are minors, hospitalized in critical and continuous surgical surveillance unit, for all surgical specialties excluding cardiac surgery. The use of central venous catheters concerns approximately 60% of the hospitalization days identified each year. To control catheter-related bacteremias, all intensive care unit patients are subjected to a service protocol since 2015, which defines a mild soap daily wash in patients without central venous catheter and a wash with Chlorhexidine in patients with central venous catheter. Successive standardized samples will be carried out on the skin of the children submissive to both types of washes during their hospitalization in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 0 to 17 years old
* Hospitalized in the pediatric surgical intensive care unit of the Necker Hospital for a duration of at least 5 days
* Patients likely to receive the 2 types of washes (mild soap and Chlorhexidine Gluconate )
* Patients subject to the service wash protocol for at least two daily washes (24 hours)

Exclusion Criteria:

* Patients not following the 2 types of washes
* Chronic skin lesions
* Refusal to participate expressed by the holders of the parental authority and/or patient
* not respecting the 24h imposed for each wash

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minors hospitalized in intensive care unit of Necker Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Cutaneous colonization | 6 months
  Number of colony-forming unit after 24 hours of culture of 3 samples : 1 hour before the wash (mild soap or 2% Chlorhexidine Gluconate), 1 to 2 hours after, and 20 to 23 hours after the wash.
Bacterial ecology | 6 months
  Macroscopic bacterial identification after Gram staining, after 24 hours of culture of 3 samples : 1 hour before the wash (mild soap or 2% Chlorhexidine Gluconate), 1 to 2 hours after, and 20 to 23 hours after the wash.
  Microbiological identification if the macroscopic appearance seems atypical.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Blanot, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Edouard Jullien, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No